CLINICAL TRIAL: NCT00970580
Title: A Phase 1b, Open-Label, Dose-Escalation Study of BIIB022 in Combination With Paclitaxel and Carboplatin in Subjects With Treatment-Naive, Stage IIIB/IV Non-Small Cell Lung Cancer
Brief Title: A Study of BIIB022 in Combination With Paclitaxel and Carboplatin in Subjects With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Therese Senta-McMillian, Clinical Team Manager, PRA International
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 212-LC-101
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2011-11

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: BIIB022; Stage IV; Taxol; Stage IIIB; Carboplatin; Paclitaxel; Non Small Cell Lung Cancer; Treatment Naive; Anti IGF1R; NSCLC; Open Label; IGF1R; Paraplatin; Cytotoxic; Mitotic Inhibitor; Taxane; Alkylating agent
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — BIIB022; Paclitaxel; Carboplatin; taxane; cixutumumab; Cytotoxins; Antimitotic Agents; Receptor Protein-Tyrosine Kinases; Alkylating Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BIIB022 in Combination with Paclitaxel and Carboplatin (Experimental): BIIB022 in Combination with Paclitaxel and Carboplatin
  Interventions: Drug: BIIB022 With Paclitaxel and Carboplatin

INTERVENTIONS:
Drug: BIIB022 With Paclitaxel and Carboplatin — Escalating doses of BIIB022 with fixed dose and schedule of paclitaxel and carboplatin
  Other Names: Taxol; Paraplatin; BIIB022; Taxane; Anti-IGF-1R; Cytotoxic; Mitotic Inhibitor; IGF-1R; Alkylating agent

SUMMARY:
The purpose of this study is to determine whether BIIB022, Paclitaxel and Carboplatin are effective in the treatment of Treatment-Naive, Stage IIIB/IV Non-Small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years old
* Treatment-naive Stage IIIB/IV Non-Small Cell Lung Cancer
* ECOG Performance Status 0 or 1

Exclusion Criteria:

* History of another primary cancer within 3 years
* Any prior or concurrent investigational or standard therapy for treatment of NSCLC
* Prior anti-IGF-1R therapy
* Unstable diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of BIIB022 in combination with paclitaxel and carboplatin | 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Resesarch Site, Los Angeles, California
  - Resesarch Site, San Diego, California
  - Resesarch Site, Denver, Colorado